CLINICAL TRIAL: NCT04724083
Title: Inflammatory Pathways and Cardiac Growth Factors Associated With Fabry Disease
Brief Title: Inflammatory Pathways and Cardiac Growth Factors Associated With Fabry Disease Cardiomyopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lysosomal and Rare Disorders Research and Treatment Center, Inc. (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-LDRTC-01
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Fabry
MeSH Terms: interventions — Environmental Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fabry Disease subjects with cardiomyopathy: Patients (males and females) with confirmed Fabry disease, with clinical cardiac involvement based on results of structural imaging (cardiac echocardiography and MRI).
  Interventions: Diagnostic Test: biomarkers
- Fabry Disease subjects without cardiomyopathy: Patients (males and females) with confirmed Fabry disease, without clinical cardiac involvement based on results of structural imaging (cardiac echocardiography and MRI).
  Interventions: Diagnostic Test: biomarkers
- Healthy control: The control group will consist of age-and gender-matched healthy individuals.
  Interventions: Diagnostic Test: biomarkers

INTERVENTIONS:
Diagnostic Test: biomarkers — new diagnostic biomarkers

SUMMARY:
In Fabry disease (FD), α-galactosidase A deficiency leads to the accumulation of globotriaosylceramide (Lyso-Gb3 and Gb3), triggering a pathologic cascade that causes progressive damage to multiple organs, including the heart. The heart is one of the organs that is very sensitive to the deficiency of α-galactosidase A. There is a subgroup of patients with significant residual α-galactosidase activity and a phenotype with primary cardiac involvement, occasionally referred as "cardiac variant." The manifestations of cardiac involvement in FD are left ventricular hypertrophy (LVH), diastolic dysfunction, microvascular angina. Cardiac hypertrophy is the most common cardiac pathology and cause of death in patients with FD. The elevation of the inflammatory markers strongly demonstrates that chronic inflammation drives the cardiovascular pathophysiology in FD. Moreover, plasma TNF, TNFR2, Il-6 specifically elevated in FD patients with cardio hypertrophy.

The chronic inflammation in combination with elevated Lyso-Gb3 further drives the FD progression even under therapy. The expression of the endothelial-cardiomyocyte growth factors will change in response to chronic inflammation during the development of cardiac hypertrophy.

This is a clinical observational study designed to identify the role of inflammatory signaling markers and secreted growth factors in the progression of cardiac pathology in FD

DETAILED DESCRIPTION:
α-Gal A catalyzes the lysosomal hydrolysis of globotriaosylceramide (Gb-3) to lactosylceramide and digalactosylceramide (Gal-Gal-Cer) to galactosylceramide (Gal-Cer). The deficiency of this enzyme leads to an accumulation of Gb-3, its metabolite, globotriaosylsphingosine (Lyso-Gb-3), and Gal-Gal-Cer in lysosomes. The deposition of Gb-3 and Lyso-Gb-3 within the myocardium is affected the cardiac function with resultant progressive cardiovascular pathology. Gb-3 accumulation was demonstrated in the cardiac valves, cardiomyocytes, nerves, and coronary arteries. At the cellular level, Gb-3 and Lyso-Gb-3 accumulation trigger a cascade of events leading to inflammation and end-stage fibrosis. In the cardiac tissue, Lyso-Gb-3 deposition is associated with increased release of inflammatory molecules and transforming growth factors. Endomyocardial biopsies show infiltration of lymphocytes and macrophages, indicating that inflammation plays a significant role in cardiac damage. Overall, accumulated data suggest that chronic inflammation leads to multisystemic FD pathology. Thus, therapeutic interventions, including enzyme replacement therapy (ERT), must be started early, before the process becomes irreversible.

The separation of reversible stages of hypertrophic cardiomyopathy from irreversible stages (1 and 2) the major challenge is the identification of an ideal "tipping point" . In patients with HCM, the elevation of the inflammatory markers NF-kB, TNF, Il-6, Il-2, TNFR1, MCP1 strongly correlates with cardiovascular pathology; however, TNF, TNFR2, and Il-6 are specifically elevated in patients with cardiac hypertrophy.

Generally, cardiac hypertrophy corresponds to the expansion of the coronary vasculature to maintain a sufficient supply of oxygen and nutrients. Thus, activation of coronary angiogenesis and fibrosis plays a vital role in cardiac vascularization and pathological hypertrophy, and tissue remodeling may cause the secretion of growth factors, VEGF, IGF-1, TGFβ, and FGF2.

NF-κB activation plays a subsequent role in the inflammatory response to cardiac dysfunction and advanced heart failure. NF-κB and TNF signaling pathways protect the heart by ischemic preconditioning; however, this protective effect depends on the concentration of TNF-α. Therefore, the appropriate concentration of TNF-α is a critical factor in the determination of the grade of cardio-pathology. Plasma circulated marker, prostaglandin D2 synthase (PTGDS), promotes cardiomyocyte survival. Integrated data from different FD studies indicates that PDGDS may be a mediator of the inflammatory process in FD. The secretion of these factors into the bloodstream activates the innate immune response. Thus, the interaction between the inflammatory pathways and cardiac vascularization is a bi-directional process. The co-coordination of these two processes and the role of ERT in influencing immune aspects of cardiac vascularization has never been explored in FD.

The purpose of this study is to identify the blood-based biomarkers for early detection of cardiac involvement and identification of different stages of hypertrophic cardiomyopathy (thickening of the heart walls) in patients with Fabry disease. The markers used to assess Fabry disease activity such as Gb3 and Lyso Gb3 will be measured. The investigators will explore different inflammatory pathways, and secreted tissue growth factors. The investigators will analyze the role of therapy, especially its timing and the activation of the immune system that relates to cardiac involvement.

The study is designed to identify the role of inflammatory signaling markers and secreted growth factors in the onset and progression of cardiac pathology in FD.

Primary objective: Identify blood-based biomarkers for early detection of cardiac involvement and identification of different stages of HCM pathology in patients with FD.

ELIGIBILITY:
Inclusion Criteria:

* approved informed consent signed by the patients,
* Confirmed diagnosis of Fabry disease based on deficient α-Gal A enzymatic activity and molecular analysis demonstrating pathogenic variants in the GLA gene
* Male and Female, ages 18-70.

Exclusion Criteria:

* Any other known genetic condition associated with HCM,
* Evidence of hepatitis B or C infections or other chronic infectious diseases,
* Pregnancy or breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (males and females) with confirmed Fabry disease, with and without clinical cardiac involvement based on results of structural imaging (cardiac echocardiography and MRI), will be included in the study. The control group will consist of age-and gender-matched healthy individuals. Cardiac involvement will be assessed using the available clinical imaging and laboratory data.
  The study will involve 30 ages-and gender-matched subjects divided into the following cohorts.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Identify blood-based biomarkers for early detection of cardiac involvement in Fabry disease | 18 months
  inflammatory markers and growth factors in blood and urine samples. Biomarkers: NF-kB, IL-2, Il-10, MCP-1,IGN-gamma, PIGF, IGF-1, TNFR, VEGF, TGF-betta, TNF-alpha, CM-CFS, Il-1a, Il-1b, Il-6.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Goker-ALpan, MD, Principal Investigator — Lysosomal and Rare Disorders Research and Treatment Center
Locations (1):
- Lysosomal and Rare disorder research and treatment center, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ivanova MM, Dao J, Friedman A, Kasaci N, Goker-Alpan O. Sex Differences in Circulating Inflammatory, Immune, and Tissue Growth Markers Associated with Fabry Disease-Related Cardiomyopathy. Cells. 2025 Feb 20;14(5):322. doi: 10.3390/cells14050322. PMID 40072051